CLINICAL TRIAL: NCT02630953
Title: Culturally and Linguistically Adapted Physical Activity Intervention for Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Dr.Bess Marcus, Professor and Chair, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Seamos Activas; 2R01NR011295 (NIH)
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Inactivity
Keywords: Physical Activity; Latinas; Spanish-language; Text-Message; English-language; Exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Original Tailored Intervention (Active Comparator): This existing empirically supported Spanish-language PA intervention, which is based on Social Cognitive Theory and the Transtheoretical Model (TTM), emphasizes behavioral strategies for increasing PA levels (goal-setting, self-monitoring, problem-solving barriers, increasing social support, self-rewards for meeting PA goals).
  Interventions: Behavioral: Original Tailored Intervention
- Enhanced Tailored Intervention (Experimental): We designed the Enhanced Tailored Intervention to build upon our previous research in order to outperform the original tailored intervention, in a cost effective, theoretically guided and data driven manner with potential for dissemination. Participants in the Enhanced Tailored Intervention will receive an interactive technology based intervention that: 1) addresses important SCT constructs for increasing PA that were not significantly changed in the original parent trial (enjoyment/outcome expectations and social support) and 2) provides greater accountability and interactivity for self-monitoring (through text messages), as requested by participants in the original parent trial.
  Interventions: Behavioral: Enhanced Tailored Intervention

INTERVENTIONS:
Behavioral: Original Tailored Intervention — The intervention includes regular mailings: weekly in month 1, biweekly in months 2 and 3, monthly in months 4 to 6, and a maintenance dose. Mailings consist of; 1) Manuals matched to the participant's current level of motivational readiness to change, based on TTM 2) Individually tailored computerized expert system feedback reports based on the participant's answers to monthly questionnaires. The computer expert system draws from a bank of over 330 messages developed from previous studies that address different levels of psychosocial and environmental factors affecting PA. 3) PA tip sheets addressing PA barriers specifically identified by Latinas in our formative research (e.g., caregiving duties, neighborhood safety).
  Arms: Original Tailored Intervention
Behavioral: Enhanced Tailored Intervention — Participants in the Enhanced Tailored arm will receive all the intervention components of the original tailored intervention, as well as: 1) additional print materials; 2) more in-depth tailored reports; and 3) text-messages. Self-monitoring was an important aspect in increasing PA in our previous trials however, participants were only asked to turn in the self-monitoring logs once a month. Based on the importance of self-monitoring and feedback from participants (R01NR011295; R01CA15994) that they wanted greater accountability and interactivity, we added a text-message component for self-monitoring.
  Arms: Enhanced Tailored Intervention

SUMMARY:
The overall goals of this renewal are to replicate the findings of Seamos Saludables in Latina women, increase the effectiveness of the intervention, and measure intervention-related changes in clinical biomarkers. We will enhance the existing intervention by incorporating participant feedback (desire for greater interactivity and accountability), further targeting Social Cognitive Theory (SCT) constructs that were not influenced overall by the original intervention yet improved amongst our most successful participants (social support, outcome expectancies), and responding to changing trends and technology use in Latinos. We will conduct a clinical trial among Latina women in California randomized to either 1) the original Seamos Saludables tailored print only intervention or 2) a theory and text messaging-enhanced interactive technology based version of the Seamos Saludables intervention. We will also measure changes in cardiovascular and metabolic biomarkers (e.g., HbA1c, and LDL) to assess potential clinical impact of the intervention.

DETAILED DESCRIPTION:
Latinos are the largest racial/ethnic minority group in the U.S., and report substantial and widening health disparities. Prevalence of type II diabetes is 60-100% higher in Latinos than in non-Latino Whites, and incidence in Latinos is projected to increase by 500% by 20503. The largest disparities are projected for Latino women (Latinas). Rates of overweight and obesity are 23% and 37% higher in Latinas than in White women respectively, and have grown faster in Mexican American women, by far the largest subgroup of Latinas, than in White women during the past decade. Given that Latinos are projected to comprise nearly one-third of the US population by 2050, this signifies a pressing public health concern in terms of costs, diminished quality of life, and lost life years. Interventions are therefore needed that are not only linguistically adapted for this population but address their specific barriers. "Mediated" intervention delivery approaches (e.g., mail, phone, or web delivered) that emphasize home-based, lifestyle activities show larger effect sizes than face-to-face approaches, are more cost-effective, are likely more sustainable, and may be particularly appropriate for Latinas, as they reduce the burden of time, childcare, and transportation, barriers commonly cited by Latinas. Thus in the previously funded parent grant (R01NR011295) we responded to PAR-07-379, "Behavioral and Social Science Research on Understanding and Reducing Health Disparities," by modifying an existing print-based mail-delivered PA intervention and adapting it specifically for Latinas in the North Eastern U.S. with low acculturation, literacy, and socioeconomic status (SES), and testing the modified intervention in a randomized controlled trial (N=266). Participants in the PA intervention arm showed significantly greater increases in at least moderate intensity activity, increasing from 1.87 min/week at baseline to 73.36 min/week at 6 months (vs. 3.02 min/week to 32.98 min/week in a contact control group). However, this is still well below the national guidelines of 150 minutes per week. This intervention therefore shows potential in promoting initial PA adoption, yet enhancements are needed to further help people achieve levels of PA that will prevent disease and reduce health disparities. The objectives of this renewal are to 1) enhance the intervention to achieve greater increases in PA, 2) assess its potential clinical impact by measuring changes in biomarkers, and 3) increase its generalizability by replicating it in Latina women, all of which would further the goal of designing an innovative behavioral intervention to promote health and prevent illness in diverse populations.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Generally healthy (If asthma, controlled high blood pressure and/or controlled type II diabetes, may be able to participate with physician consent)
* Sedentary (Less than 60 minutes per week of moderate or vigorous physical activity)
* Hispanic or Latina (self-identified)
* Must be able to read and write in English or Spanish fluently
* 18 - 65 years of age
* Planning on living in the area for the next 12 months
* Own a cell phone capable of sending and receiving text messages

Exclusion Criteria:

* BMI greater than 45
* Not able to walk continuously for 30 minutes/limited ability to complete daily activity or ability to exercise
* Exercise is against advice of doctor
* Current or planned pregnancy
* Heart disease/treatment
* Heart murmur
* Angina/chest pain or Angina/chest pain with exertion
* Palpitations
* Stroke/Transient Ischemic Attacks
* Peripheral Vascular Disease
* Type I Diabetes
* Uncontrolled Type II Diabetes
* Chronic Infectious Disease - HIV, Hepatitis
* Chronic liver disease
* Cystic Fibrosis
* Abnormal EKG on last EKG performed
* Emphysema, Chronic bronchitis, Chronic Obstructive Pulmonary Disease
* Seizure in past year
* Surgery in past year on heart, lung, joint, orthopedic surgery
* Surgery pending in next year on lung, joint, orthopedic surgery
* Unusual/concerning shortness of breath
* Asthma (may be able to participate with physician consent)
* High blood pressure/high blood pressure medication (may be able to participate with physician consent)
* Use of beta blockers
* Abnormal Medical Stress Test
* Musculoskeletal problems
* Fainting/dizziness more than 3 times in past year OR interferes with daily activities OR causes loss of balance
* Cancer treatment in past 3 months
* Hospitalized for psychiatric disorder in past 3 years or suicidal

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bess H Marcus, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Larsen B, Gilmer T, Pekmezi D, Hartman SJ, Benitez T, Rabin B, Marcus BH, Mendoza-Vasconez AS, Groessl EJ. Cost effectiveness of a technology-enhanced physical activity intervention for Latinas. Transl Behav Med. 2023 Sep 12;13(9):675-682. doi: 10.1093/tbm/ibad021. PMID 37208924
- [Derived] Marcus BH, Dunsiger S, Pekmezi D, Benitez T, Larsen B, Meyer D. Physical activity outcomes from a randomized trial of a theory- and technology-enhanced intervention for Latinas: the Seamos Activas II study. J Behav Med. 2022 Feb;45(1):1-13. doi: 10.1007/s10865-021-00246-6. Epub 2021 Aug 11. PMID 34379236

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants attended an in-person orientation session where they received information about the study, had measures of height, weight, and self-reported PA taken to confirm eligibility. During a second visit, participants were measured (e.g, hip and waist circumference)) and given an ActiGraph GT3X+ accelerometer. After one week of continuous accelerometer wear, participants returned for their baseline visit where they completed questionnaires, had blood draws, then were randomized/
Period: 6 Month Assessment
Arm/Group | Original Tailored Intervention | Enhanced Tailored Intervention
Started | 97 | 102
Completed | 83 | 70
Not Completed | 14 | 32
Period: 12 Month Assessment
Arm/Group | Original Tailored Intervention | Enhanced Tailored Intervention
Started | 97 | 102
Completed | 73 | 64
Not Completed | 24 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Original Tailored Intervention | Enhanced Tailored Intervention | Total
Number analyzed (Participants) | 97 | 102 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.14 (9.57) | 43.55 (10.63) | 43.80 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 102 | 199
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 97 | 102 | 199
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 45 | 47 | 92
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 44 | 52 | 96
Region of Enrollment [Number; unit: participants]
  United States | 97 | 102 | 199
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.79 (5.19) | 30.50 (9.31) | 30.64 (7.56)
Self Reported Min/Week MVPA [Mean (Standard Deviation); unit: minutes/week] | 10.51 (19.47) | 14.33 (25.06) | 12.47 (22.54)
Objectively Measured Min/Week MVPA [Mean (Standard Deviation); unit: minutes/week] | 45.72 (70.93) | 33.61 (71.29) | 39.51 (71.20)

OUTCOME MEASURES:

1. Primary Outcome: Change in Accelerometer Measured Moderate to Vigorous PA (MVPA) by the Actigraph GT3X+
Description: Participants will wear an Actigraph GT3X+ accelerometer, which measures movement and intensity of activity and has been validated against heart rate telemetry and total energy expenditure.
Time Frame: Baseline, 6 months and 12 months
Population: Analysis was completed on the ITT sample
Measure: Median (Inter-Quartile Range); unit: minutes/week
Arm/Group | Original Tailored Intervention | Enhanced Tailored Intervention
Number analyzed (Participants) | 97 | 102
minutes/week
  Baseline | 10 [0 to 68.50] | 0 [0 to 38]
  6 Months | 36 [0 to 109.75] | 28 [0 to 98.50]
  12 Months | 36 [0 to 127] | 40 [0 to 110]
Statistical Analysis 1: Comparison: Original Tailored Intervention vs Enhanced Tailored Intervention; Using a series of quantile regression models with bootstrapped standard errors (10,000 replications) we examined the potential treatment effects on MVPA at follow-ups, controlling for baseline. Quantile regression models the median outcome instead of the mean, and are appropriate when data is skewed (as was the case in both self-reported and objectively measured MVPA); Test type: Superiority; p = 0.24, quantile regression — Significance level was set at .05 a priori; Bootstrapped standard errors (10,000 replications); Median Difference (Final Values) = -6.22, 95% CI 2-sided [-41.15 to 28.70]

2. Secondary Outcome: Change in Total Weekly Minutes of Physical Activity as Measured by the 7-Day PAR (Physical Activity Recall), From Baseline to 6-months and 12-months.
Description: The 7-Day PAR is an interviewer administered instrument that uses multiple strategies for increasing accuracy of participant recall regarding many types of activities such as time spent sleeping and moderate, hard, and very hard intensity activities. The 7-Day PAR is used across many studies assessing physical activity and has consistently demonstrated acceptable reliability, internal consistency, and congruent validity with other objective measures of activity levels.
Time Frame: Baseline, 6 months and 12 months
Population: Analysis was completed on the ITT sample
Measure: Median (Inter-Quartile Range); unit: minutes/week
Arm/Group | Original Tailored Intervention | Enhanced Tailored Intervention
Number analyzed (Participants) | 97 | 102
minutes/week
  Baseline | 0 [0 to 15] | 0 [0 to 20]
  6 Months | 100 [30 to 172] | 110 [66 to 175]
  12 Months | 100 [43.50 to 183] | 130 [45 to 195]
Statistical Analysis 1: Comparison: Original Tailored Intervention vs Enhanced Tailored Intervention; Using a series of quantile regression models with bootstrapped standard errors (10,000 replications) we examined the potential treatment effects on MVPA at follow-up, controlling for baseline; Test type: Superiority; p = 0.73, quantile regression — Significance was set at .05 a priori; Median Difference (Final Values) = 7.5, 95% CI 2-sided [-32.37 to 47.37]

3. Secondary Outcome: Changes in Cardiovascular and Metabolic Biomarkers (e.g., HbA1c, and LDL)
Description: Blood samples will be collected at the baseline and 6-month clinic visits. Specifically, low-density lipoprotein cholesterol (LDL), hemoglobin A1C (HbA1c), and blood pressure will be measured. These assays will be collected by personnel at the UCSD NIH-funded Clinical and Translational Research Institute (CTRI).
Time Frame: Baseline, 6 months
Population: A subset of the full sample completed biomarker analysis at baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Original Tailored Intervention | Enhanced Tailored Intervention
Number analyzed (Participants) | 78 | 75
percentage
  Baseline A1c | 5.36 (0.38) | 5.43 (0.83)
  6 Month A1c | 5.35 (0.43) | 5.29 (0.27)
Statistical Analysis 1: Comparison: Original Tailored Intervention vs Enhanced Tailored Intervention; Using a series of generalized linear models with identity link, we examined treatment effects on biomarkers at 6 months controlling for baseline and potential confounders; Test type: Superiority; p > .06, Regression, Linear — Significance level set at .05 a priori; Mean Difference (Net) = -.06, Standard Error of Mean .035

4. Secondary Outcome: Changes in Cholesterol
Description: Blood samples will be collected at the baseline and 6-month clinic visits. Specifically, low-density lipoprotein cholesterol (LDL) will be measured. These assays will be collected by personnel at the UCSD NIH-funded Clinical and Translational Research Institute (CTRI).
Time Frame: Baseline, 6 months
Population: A subset of the full sample completed biomarker analysis at baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Original Tailored Intervention | Enhanced Tailored Intervention
Number analyzed (Participants) | 78 | 75
mg/dL
  Baseline Cholesterol | 188.65 (31.70) | 192.00 (37.29)
  6 Month Cholesterol | 188.09 (31.17) | 185.42 (38.42)
  Baseline HDL | 51.13 (12.54) | 52.28 (54.13)
  6 Month HDL | 53.44 (12.38) | 54.13 (13.50)
  Baseline LDL | 104.80 (26.56) | 109.75 (30.94)
  6 Month LDL | 109.41 (28.43) | 107.71 (31.05)

5. Secondary Outcome: Changes in Triglycerides
Description: Blood samples will be collected at the baseline and 6-month clinic visits.
Time Frame: Baseline, 6 months
Population: A subset of the full sample completed biomarker analysis at baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Original Tailored Intervention | Enhanced Tailored Intervention
Number analyzed (Participants) | 78 | 75
mg/dL
  Baseline Triglycerides | 166.58 (101.60) | 149.88 (117.94)
  6 Month Triglycerides | 133.91 (90.98) | 117.94 (57.40)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Original Tailored Intervention | Enhanced Tailored Intervention
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/102
Other Adverse Events (participants affected / at risk) | 5/97 | 10/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Tailored Intervention (N=97) | Enhanced Tailored Intervention (N=102)
Toe Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Participant reported feeling pain in her big toe. She stated that the pain is due to a bunion on her foot that she has had for the past 20 years. She sees her physician regularly and they have not advised her to discontinue physical activity.
Infected Bladder (Renal and urinary disorders) | 0 (0) | 1 (1) — Participant stating that she just had surgery for an infected bladder. Her physician had instructed her to do no extraneous physical activity until further notice. Participant was put on medical hold until she could receive clearance.
Hip Pain and Rash (General disorders) | 0 (0) | 1 (1) — Participant reporting that she had a rash on her leg and minor pain in her left hip but that she no longer feels any pain.
Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — 1. Participant had a pain in her leg when playing basketball and Zumba. 2. Participant's legs were bothering her with pain after 1 mile of fast walking.
Heel and Back Pain (General disorders) | 1 (1) | 0 (0) — Participant reported pain in her heels which continued through the night and began to bother her back. She stated that she suffers from ingrown toenails and speculated that this condition may exacerbate the foot pain.
Knee Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — 1. Participant reported that she twisted her knee while standing in her kitchen. She stated that this injury was not related to the study. 2. We received a completed adverse event form reporting that the participant has had knee pain
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Participant reported having lumbar spinal stenosis. The participant is confident that the pain/sciatica was not brought on by the exercise in the study and says the walking has actually been helpful.
Foot Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — We received a completed adverse event from this participant stating pain in her foot.
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — 1. We received a completed adverse event from this participant stating that she has knee pain. 2. We received a completed adverse event form reporting that the participant had pain in her right knee what she ran.
Leg Injury (General disorders) | 1 (1) | 0 (0) — We received a completed adverse event form reporting that the participant hurt her leg when standing on top of a gallon jug and that she scratched and bruised her leg.
Breast Biopsy (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Participant had a minor biopsy to remove a small sample from her left breast.
Stroke (unrelated to study) (Cardiac disorders) | 0 (0) | 1 (1) — Participant informed our staff member via phone that her daughter in the study had suffered a stroke last month while at school and thus she felt like it was necessary for her and her daughter withdraw from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT02630953/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT02630953/SAP_001.pdf